CLINICAL TRIAL: NCT02034981
Title: AcSé CRIZOTINIB : Secured Access to Crizotinib for Patients With Tumors Harboring a Genomic Alteration on One of the Biological Targets of the Drug.
Brief Title: Phase 2 Study Assessing Efficacy and Safety of Crizotinib in Patients Harboring an Alteration on ALK, MET or ROS1
Acronym: AcSé
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: National Cancer Institute, France (Other Government); Fondation ARC (Other); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UC-0105/1303; 2013-000885-13 (EudraCT Number)
Record Dates: First submitted 2013-10-16; First posted 2014-01-14 (Estimated); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Hematologic Cancers; Solid Tumors; Metastatic Cancer
Keywords: metastatic or unresectable locally advanced malignancies.; genomic alterations.; biological crizotinib targets (ALK, MET, ROS1, RON, AXL).
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Crizotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CRIZOTINIB (Experimental): All eligible patients entering the study will receive oral crizotinib as monotherapy
  Interventions: Drug: Crizotinib

INTERVENTIONS:
Drug: Crizotinib — Patients will receive oral crizotinib, daily continuously, until progression or unacceptable toxicity develops.
  -250 mg twice daily for adults ≥ 18 years of age
  * 280 mg/m² twice daily for children and adolescents aged from 1 to 17 (except ALCL).
  * 165 mg/m² twice daily for ALCL patients aged from 1 to 17.
  Other Names: XALKORI

SUMMARY:
This is a biology driven, trans-tumoral, multicentric phase II trial assessing the efficacy and the safety of the targeted agent crizotinib as a monotherapy in 23 cohorts of patients with identified activating molecular alterations in the crizotinib target genes. A cohort is defined by a pathology and a crizotinib-target alteration (eg gastric cancer with MET amplification).

For each cohort a two-stage design will be implemented. In the situation where expected accrual allows for a sufficient number of patients to be accrued, the alpha and beta errors will be fixed at 10%. However, in very rare diseases, such as inflammatory myofibroblastic tumor (IMT), neuroblastoma, glioblastoma, and rhabdomyosarcoma (RMS), it is anticipated that the target number may not be achievable in a reasonable timeframe; for these cohorts, the alpha and beta errors will be fixed at 15%. Consequently three different statistical designs will be a priori considered according to the expected response rate and incidence.

DETAILED DESCRIPTION:
Twenty cohorts are identified, a cohort being defined as [one pathology, one target alteration] such as [gastric cancer with MET amplification (6%)].

One cohort will be dedicated to miscellaneous, very rare pediatric diseases identified through INCa platforms or pan-genome programs (e.g. MOSKIDO, IGR) and will recruit up to 10 patients.

Two cohorts will be dedicated to a couple of diseases harbouring at least one specific alteration in one crizotinib target, same or different from those listed above, e.g. in AXL gene, arising from pan-genome trials.

1. ALCL, adults and children, ALK-translocated
2. Colorectal cancer, adults, ALK-translocated
3. Colorectal cancer, adults, MET amplified
4. Colorectal cancer, adults, MET mutated
5. NSCLC, adults, MET amplified
6. NSCLC, adults, ROS1-translocated
7. Breast cancer, adults, ALK-translocated
8. Gastric cancer, adults, MET amplified
9. Cholangiocarcinoma, adults, ROS1-translocated
10. Ovarian cancer, adults, MET amplified
11. Clear cell renal cell carcinoma, adults, ALK-translocated
12. Clear cell renal cell carcinoma, adults, ALK-amplified
13. Papillary renal cell carcinoma, adults, MET mutated (+ MET amplified)
14. Hepatocarcinoma, adults, MET amplified
15. Neuroblastoma, adults and children, ALK-amplified + ALK mutated
16. IMT, adults and children, ALK-translocated
17. Rhabdomyosarcoma (alveolar and embryonal), adults and children, ALK-amplified
18. Glioblastoma, adults, MET amplified. This cohort will only be open after amendment
19. Anaplastic thyroid cancer, adults, ALK mutated
20. Thyroid cancer (follicular + medullary + papillary), adults, MET mutated
21. Miscellaneous rare pediatric diseases associated to at least one specific alteration in one crizotinib target, same or different from those listed above
22. One another pathology associated to at least one specific alteration in one crizotinib target, same or different from those listed above.
23. One another pathology associated to at least one specific alteration in one crizotinib target, same or different from those listed above.

ELIGIBILITY:
Inclusion:

* Male and female ≥ 1 year of age
* unresectable locally advanced or metastatic malignant tumor of any histological type (but NSCLC with an ALK translocation) and not amenable to any other validated therapeutic option. ( for pediatrics a relapse after a first well-conducted standard treatment or a situation without any standard treatment and a survival <10%).
* one proven specific alterations among ALK, MET, RON and ROS1 genes determined on the primary and/or the metastatic lesion
* Measurable disease according to RECIST 1.1
* For patients with primary cerebral tumors (adults or children), measurable disease defined by bi-dimensional measurements : two perpendicular diameters of at least 10 mm on CT or MRI scan, outside of a previously radiated field within the last 3 months, to observe pseudoprogression
* hematologic function (ANC ≥ 1.0x10⁹/L, platelets ≥ 75x10⁹/L, platelets ≥ 50x10⁹/L for ALCL with bone marrow involved ; platelets ≥ 100x10⁹/L for primary or secondary cerebral tumors; Hb ≥ 8g/L), renal function (creat cl ≥ 50 mL/min Cockcroft and Gault) and hepatic function (serum bilirubin ≤ 1.5x ULN unless due to Gilbert's syndrome ; ASAT and ALAT ≤ 5x ULN if liver metastasis or ≤ 3x ULN if liver metastasis with advanced fibrosis (FibroTest>0.48) or ≤ 3x ULN without liver metastasis)
* normal values for calcium, magnesium and potassium levels
* able to swallow and retain oral medication
* ECOG Performance Status of 0 to 2, or Karnofsky scale > 50 % or Lansky Play scale (< 12 years) > 50%, (for CNS tumors, the neurological deficiency due to the disease itself)
* Life expectancy ≥ 3 months

Exclusion :

* NSCLC patients ALK translocations
* Patient eligible for a clinical trial with an anticancer drug (including crizotinib) targeting the same molecular alteration open to accrual in France.
* alteration limited to an overexpression of ALK, MET, RON, ROS1 or any other crizotinib-target. Only patients with ALCL are eligible if ALK is positive by immunohistochemistry
* Patients with primary or secondary central nervous system disease
* Previous treatment with crizotinib
* Major surgery or tumor embolization within 4 weeks and minor surgery within 2 weeks prior to the initiation of the study drug. Brain surgery is excluded within 4 weeks prior to starting crizotinib for primary or secondary cerebral tumors
* Patients with other concurrent severe and/or uncontrolled medical disease which could compromise participation in the study, such as, but not limited to :

  * Within the 3 months prior to starting study treatment: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, or cerebrovascular accident including transient ischemic attack
  * Ongoing congestive heart failure
  * Congenital long QT syndrome
  * Heart rate ≤ 45 beats/minute
  * Ongoing cardiac dysrhythmias of NCI CTCAE Grade ≥2, uncontrolled atrial fibrillation of any grade, or with QTcF interval >470 msec
  * For patients with a cerebral disease (primary or secondary) : uncontrolled hypertension [defined as SBP of ≥ 140 mmHg or DBP of ≥ 90mmHg]
  * extensive disseminated/bilateral or known presence of Grade 3 or 4 interstitial fibrosis or interstitial lung disease, including pneumonitis, hypersensitivity pneumonitis, interstitial pneumonia, interstitial lung disease, obliterative bronchiolitis, and pulmonary fibrosis, but not prior radiation pneumonitis
  * Spinal cord compression unless treated with the patient attaining good pain control and stable or recovered neurologic function
  * Carcinomatous meningitis or leptomeningeal disease
  * HIV-positive, active hepatitis A, B or C, or latent hepatitis B or C, or any other uncontrolled infection
  * Other severe acute or chronic medical or psychiatric conditions, or end stage renal disease on hemodialysis or laboratory abnormalities
  * For patients with a cerebral disease, detection on the MRI or the CTscan of a real arteriovenous malformation, or an untreated intracranial aneurysm, or a cavernous angioma, or an amyloid angiopathy, or any new or significant (≥ grade 2) intratumoral bleeding other than microbleeds on T2* weighted MRI in the previous 14 days before treatment initiation, or a recent and untreated subdural effusion.
* Patients using non-substitutable drugs that are potent CYP3A4 inhibitors, or potent CYP3A4 inducers
* Patients using non-substitutable drugs that are CYP3A4 substrates with narrow therapeutic indices
* Patients with cerebral disease using anti-platelet drugs or anticoagulant agents are not eligible if those treatments can not be stopped 7 days before day1.
* Patients with altered mental status or with psychological, familial, sociological or geographical condition potentially hampering compliance
* Individual deprived of liberty or placed under the authority of a tutor.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2023-12-06 (Actual)

PRIMARY OUTCOMES:
The efficacy of crizotinib as a single agent across diverse type of tumors guided by the presence of identified activating molecular alterations in the crizotinib target genes, per cohort, per pathology, and per target. | Determined after 8 weeks (2 cycles) of treatment
  Anti-tumor activity of crizotinib, as the primary objective of the trial, will be carried out by the determination of the objective response assessed in each cohort defined by a pathology associated with a crizotinib target alteration.
  The objective response is defined as either a complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria.
  The objective response after 2 cycles (8 weeks) will be reported to define a success in the 2-stage design.

SECONDARY OUTCOMES:
The safety profile of crizotinib. | Safety profile will be assessed during the whole treatment period (6 months expected in average) followed by a 2-year post-treatment follow-up period, and reported during the visits scheduled by the study flow chart
  Toxicities will be assessed by clinical and paraclinical examinations at every scheduled visit during the whole treatment period and the post-treatment follow-up period (around 2.5 years) This study will use the International Common Terminology Criteria for Adverse Events (CTCAE), version 4.0, for adverse event reporting.
Disease control rate | After 8 weeks (2 cycles) and 16 weeks (4 cycles) of treatment
  Disease Control Rate will be the percentage of patients with a CR, PR or Stable Disease (SD) according to RECIST at the end of cycle 2 (8 weeks) and at the end of cycle 4 (16 weeks) in the group of patients evaluable for response
response duration | interval between the objective response (CR or PR) and time of progression, recurrence or death
  Response duration will be the time interval between the date that the criteria of CR/PR (whichever is first recorded) are met for the first time and the first date of documented re-appearance of the disease (recurrence, progression or death). If neither event has been observed, then the patient is censored at the date of the last follow up examination.
Progression-free survival | from registration until time of disease progression or death
  Progression-free survival will be the time interval between the date of registration and the day of first documented sign of disease progression (first day when RECIST criteria of progression are met) or day of death whatever the cause (events). If neither event has been observed, then the patient is censored at the date of the last follow up examination.
Overall survival | from registration until date of death
  Overall survival will be the time interval between the date of registration and the date of death, whatever the cause of death. Patients still alive at follow-up are censored at the date of last follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Gilles VASSAL, Principal Investigator — Gustave Roussy, Villejuif
Locations (1):
- Gustave Roussy, Villejuif, Île-de-France Region, France

REFERENCES:
- [Derived] Brugieres L, Cozic N, Houot R, Rigaud C, Sibon D, Arfi-Rouche J, Bories P, Cottereau AS, Delmer A, Ducassou S, Garnier N, Lamant L, Leruste A, Millot F, Moalla S, Morschhauser F, Nolla M, Pagnier A, Reguerre Y, Renaud L, Schmitt A, Simonin M, Verschuur A, Hoog Labouret N, Mahier Ait Oukhatar C, Vassal G. Efficacy and safety of crizotinib in ALK-positive systemic anaplastic large-cell lymphoma in children, adolescents, and adult patients: results of the French AcSe-crizotinib trial. Eur J Cancer. 2023 Sep;191:112984. doi: 10.1016/j.ejca.2023.112984. Epub 2023 Jul 17. PMID 37549532
- [Derived] Aparicio T, Cozic N, de la Fouchardiere C, Meriaux E, Plaza J, Mineur L, Guimbaud R, Samalin E, Mary F, Lecomte T, Gomez-Roca C, Haineaux PA, Gratet A, Selves J, Menu Y, Colignon N, Johnson L, Legrand F, Vassal G. The Activity of Crizotinib in Chemo-Refractory MET-Amplified Esophageal and Gastric Adenocarcinomas: Results from the AcSe-Crizotinib Program. Target Oncol. 2021 May;16(3):381-388. doi: 10.1007/s11523-021-00811-8. Epub 2021 Apr 13. PMID 33847874
- [Derived] Moro-Sibilot D, Cozic N, Perol M, Mazieres J, Otto J, Souquet PJ, Bahleda R, Wislez M, Zalcman G, Guibert SD, Barlesi F, Mennecier B, Monnet I, Sabatier R, Bota S, Dubos C, Verriele V, Haddad V, Ferretti G, Cortot A, De Fraipont F, Jimenez M, Hoog-Labouret N, Vassal G. Crizotinib in c-MET- or ROS1-positive NSCLC: results of the AcSe phase II trial. Ann Oncol. 2019 Dec 1;30(12):1985-1991. doi: 10.1093/annonc/mdz407. PMID 31584608